CLINICAL TRIAL: NCT05734703
Title: Skin Rejuvenation Using Topical Hemp-based Extract and Other Nutraceuticals
Brief Title: Skin Rejuvenation With Topical Extract and Other Nutraceuticals
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Life Care Planners, LLC (Other)
Responsible Party: Principal Investigator, Gregory L Smith, MD, MPH, Principal Investigaor, Medical Life Care Planners, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Skin Antiaging Effects
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Wrinkle; Spot Pigmented; Lines Skin
Keywords: hemp extract; caffeine; resveratrol; thyme
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: One group of 25 adults aged 50 or over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Standard Topical Daily Dose (Experimental): Only one arm in the study. Subjects treated with the topical daily for 90 days. The comparison will be 'before' and 'after' treatment skin biopsy results.
  Interventions: Drug: Nutraceutical Topical

INTERVENTIONS:
Drug: Nutraceutical Topical — Once daily application of the topical nutraceutical to two by two inch area of skin for 90 days.

SUMMARY:
Hemp extract has been shown in several pre-clinical and clinical studies to have anti-aging effects on the skin through anti-oxidant and anti-inflammatory effects, in addition resveratrol, thyme and caffeine have been shown to have anti-aging effects related to fibrillar collagen production and extracellular matrix production in the dermis.

A combination of these four ingredients will be used in a vehicle of fermented medium chain triglyceride oil and skin shave biopsies will be taken before and after 90 days use of the topical to look for objective evidence of anti-aging effects in the dermis and epidermis.

DETAILED DESCRIPTION:
The study is a case series of 25 adults over age 50 identified through social media outreach in the Tampa Bay area. Each subject will be given a topical serum and advised to apply it once daily to the specific two by two inch area of skin under study (forearm or back of the neck). The serum will be comprised of hemp-extract, resveratrol, caffeine, thyme oil and fermented medium chain triglyceride as a vehicle. The skin anti-aging serum is expected to contain hemp-extract 5%, caffeine 2%, Thyme essential oil 2% and resveratrol 0.5%. The subjects will use the test formulation for 90 days. The subjects will jhave shaved skin biopsies taken on either the forearm or back of the neck. The biopsies will be done on day zero and on day 90.

None of the subjects are currently using anti-aging therapies. No other anti-aging therapy will be used during the 90 days of the research.

The subjects will be advised to apply a thin layer of the serum once each night at bedtime. To the area of skin under study (forearm or back of the neck). The one-ounce bottle of serum is expected to last for the entire 90 days of the study. The subjects will be reminded each day via text messaging to use the product and each subject will be required to text back that the daily treatment has been applied.

The 'before and after' shaved biopsies will be independently evaluated by Dr. Michael Morgan, board certified Dermatopathologist at KorPath, Inc. He will perform hematoxylin and eosin (H&E) staining, for histological analysis for morphology of the dermis and epidermis and histochemical staining for collagen and matrix analysis.

The subjects will be independently clinically evaluated by Dr. Kathy Anderson, board certified Dermatologist. She will determine "before and after" skin wrinkling scores using standard recognized metrics.

Each subject will have a diary app added to their smart phones to document daily use and potential adverse effects.

The results will be statistically evaluated with a standard for comparison. Study results with a p-value less than 0.05 will be determined to be statistically significant and the result will be evaluated for efficiency compared to generally recognized therapies

. The study will be prepared in standard fashion and submitted to recognized peer-review medical journals.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or over
* Glogau Wrinkle Severity Scale of either 3 or 4 on the area to be biopsied.
* Not on current anti-aging therapies used as an ingredient in the study topical.

Exclusion Criteria:

* Under age 50
* Glogau Wrinkle Severity Scale of either 1 or 2 on the area to be biopsied.
* Currently using anti-aging therapies used as an ingredient in the study topical.
* Contraindication to performing skin shave biopsies in the area to be biopsied.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
dermal-epidermal juncton flattening | 90 days
  Histologic appearance of dermal-epidermal flattening on 'before' and 'after' skin biopsies.
elastic fiber attenuation | 90 days
  Histologic appearance of elastic fiber attenuation in the dermis on 'before' and 'after' skin biopsies.
denisty of collagen fiber network | 90 days
  Histologic appearance of the density of the collagen fibers on 'before' and 'after' skin biopsies.

SECONDARY OUTCOMES:
Glogau System: Wrinkle Severity Ranking | 90 days
  Glogau System: Wrinkle Severity Ranking score from 1-4 on 'before' and 'after' dermatologist physical examination of treated area
Modified Fitzpatrick Wrinkle Scale | 90 days
  Modified Fitzpatrick Wrinkle Scale from class 0-2.5 on 'before' and 'after' dermatologist physical examination of treated area

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Smith, MD, Principal Investigator — Nex Therapeutics, LLC
Locations (1):
- Laser Scalp and Hair Center, Clearwater, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Caverzan J, Mussi L, Sufi B, Padovani G, Nazato L, Camargo FB Junior, Magalhaes WV, Di Stasi LC. A new phytocosmetic preparation from Thymus vulgaris stimulates adipogenesis and controls skin aging process: In vitro studies and topical effects in a double-blind placebo-controlled clinical trial. J Cosmet Dermatol. 2021 Jul;20(7):2190-2202. doi: 10.1111/jocd.13818. Epub 2020 Nov 10. PMID 33169920
- [Result] Costa EF, Magalhaes WV, Di Stasi LC. Recent Advances in Herbal-Derived Products with Skin Anti-Aging Properties and Cosmetic Applications. Molecules. 2022 Nov 3;27(21):7518. doi: 10.3390/molecules27217518. PMID 36364354
- [Result] Few J, Lee MJ, Semersky A, Mariscal E, Vachon G. A Single-Center Study Evaluating the Effects of a Novel Retinol and Cannabidiol Combination Topical on Facial Skin. Aesthet Surg J Open Forum. 2022 Jan 27;4:ojac002. doi: 10.1093/asjof/ojac002. eCollection 2022. PMID 35274096